CLINICAL TRIAL: NCT07082400
Title: Screening and Phenotyping of Pulmonary Hypertension in Heart Failure With Preserved Ejection Fraction .
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Sayed, assistant lecturer chest department faculty of medicine Sohag University, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Soh-Med-25-6--3MD
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: right heart catheter — measurement of hemodynamics of pulmonary circulation in patients diagnosed with heart failure with preserved ejection fraction

SUMMARY:
Left-sided heart failure (HF) is known to cause pulmonary hypertension (PH), but the development and severity of PH in HF is highly variable, and contributing factors are not fully understood. Pulmonary hypertension (PH) due to left heart disease (PH-LHD) is a growing health problem with high morbidity and mortality . PH-LHD is the most frequent subset of PH, resulting from left ventricular (LV) dysfunction (systolic and/or diastolic) and/or valvular heart disease (VHD) . Although initial studies focused on patients with reduced left ventricular ejection fraction (EF) , early isolated case reports and more recent case series have shown that PH can occur in heart failure with preserved ejection fraction (HFpEF). There is now growing appreciation that PH is common and may be severe in elderly patients with HFpEF . However, the true prevalence and severity of PH in HFpEF from the general community remain unknown. Previous studies were limited by selection bias, and population-based data have, to date, been lacking. Common to left ventricular failure regardless of EF, increased left-sided filling pressure leads to pulmonary venous hypertension (HTN) and post-capillary PH. In the presence of preserved systolic function, the development of pulmonary venous HTN is associated with the severity of left ventricular diastolic dysfunction, as has been shown in patients with aortic stenosis and normal EF. Beyond this post-capillary contribution to PH, a reactive increase in pulmonary arterial tone or intrinsic arterial remodeling can result in a superimposed pre-capillary component of pulmonary arterial HTN. This has been shown to occur in patients with mitral stenosis and HF with reduced EF. In HFpEF without valvular disease, however, the relative contributions of these pre- and post-capillary components to PH are unclear. Pulmonary arterial compliance (CPA) is a predictor of prognosis in patients with SHF, irrespective of pulmonary vascular resistance (PVR).Recently, at the fifth World Symposium on Pulmonary Hypertension in Nice, France, in 2013, two subsets of PH-LHD (post-capillary PH) were defined as isolated post-capillary PH (Ipc-PH; diastolic pulmonary vascular pressure gradient [DPG] < 7 mm Hg, previously labeled as "passive" PH-LHD) and combined pre- and post-capillary PH (Cpc-PH; DPG ≥ 7 mm Hg, previously labeled as "out-of-proportion" or "reactive" PH-LHD, because of pulmonary pressures higher than expected from increased pulmonary artery wedge pressure (PAWP). HF therapies such as β-blockers, angiotensin-converting enzyme inhibitors, angiotensin receptor blockers, and spironolactone improve LV function and reduce LV filling pressures, but have not been convincingly shown to improve RV function in humans. In contrast, pulmonary vasodilators that have been approved for the treatment of pulmonary arterial hypertension (PAH) have never demonstrated a benefit in HF populations, including recent randomized trials . There are Diagnostic Dilemmas as diastolic heart failure causing pulmonary hypertension and pulmonary hypertension causing diastolic dysfunction. Chronic right ventricular pressure overload can affect left ventricular diastolic function in several ways. Left ventricular relaxation is under the triple control of load, myocardial properties, and the uniformity of load in space and time .18 In chronic right ventricular pressure overload, the load on the intraventricular septum is dramatically increased and as it hypertrophies, the myocardial properties of the septum are altered. The motion of the intraventricular septum in systole and diastole is asynchronous. All these factors could contribute to impairment in global left ventricular relaxation. In Doppler echocardiographic studies of IPAH, impaired relaxation with decreased E/A ratio and increased isovolumic relaxation time and deceleration time have been consistently reported . While patients must have normal PCWP to be diagnosed with IPAH, there is considerable evidence that chronic right ventricular pressure overload can cause reduced left ventricular compliance. The external forces affecting the LV-EDPVR include right ventricular pressure and pericardial pressure.19_20 The effect of right ventricular pressures on the LV-EDPVR is termed "ventricular interdependence" and is accentuated in the presence of an intact pericardium . These effects were also apparent in chronic right ventricular pressure overload, but a decrease in myocardial compliance (as assessed by the stress-strain relationship) was also seen.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with diastolic heart failure through The H2FPEF score and suspected pulmonary hypertension

Exclusion Criteria:

* Heart Failure with reduced ejection fraction .
* Severe lung diseases as a comborbid condition ,such as COPD (GOLD) class 4 , severe interstitial lung disease.
* Chronic thromboembolic PH .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
mean pulmonary arterial pressure | 1 year
  through right heart catheter

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Maron BA, Bortman G, De Marco T, Huston JH, Lang IM, Rosenkranz SH, Vachiery JL, Tedford RJ. Pulmonary hypertension associated with left heart disease. Eur Respir J. 2024 Oct 31;64(4):2401344. doi: 10.1183/13993003.01344-2024. Print 2024 Oct. PMID 39209478
- [Background] Wissmuller M, Dohr J, Adler J, Ochs L, Tichelbacker T, Hohmann C, Baldus S, Rosenkranz S. Pulmonary hypertension associated with left heart disease. Herz. 2023 Aug;48(4):266-273. doi: 10.1007/s00059-023-05189-z. Epub 2023 Jun 8. PMID 37289211
- [Background] Madonna R, Biondi F, Ghelardoni S, D'Alleva A, Quarta S, Massaro M. Pulmonary hypertension associated to left heart disease: Phenotypes and treatment. Eur J Intern Med. 2024 Nov;129:1-15. doi: 10.1016/j.ejim.2024.07.030. Epub 2024 Aug 1. PMID 39095300
- [Background] Redfield MM, Borlaug BA. Heart Failure With Preserved Ejection Fraction: A Review. JAMA. 2023 Mar 14;329(10):827-838. doi: 10.1001/jama.2023.2020. PMID 36917048